CLINICAL TRIAL: NCT01643343
Title: Measurement of Joint Attention Fluency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Vista School (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: 33060
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Autism Spectrum Disorders; Autism
Keywords: autism spectrum disorders; autism; joint attention; imitation; fluency
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Typically Developing: Typically developing toddler volunteers between the ages of 8 months and 3 years
- Autism: Children between the ages of 8 months and 6 years with a diagnosis of an autism spectrum disorder

SUMMARY:
The purpose of this research is to study joint attention. Joint attention plays a critical role in social and language development in children with and without autism. Joint attention is the shared attention between a child and another person. This study seeks to set a standard benchmark of frequency scores for joint attention. Finding a rate of engaging in joint attention behavior would offer a benchmark for all researchers and practitioners working with learners with and without autism.

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder

Exclusion Criteria:

* hearing or vision problems
* behaviors that are a danger to self or others

Ages: 8 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The Vista School, Hershey, Pennsylvania, United States